CLINICAL TRIAL: NCT07226219
Title: Pilot Trial of Stimulant Treatment to Address Attention and Executive Deficits Among Children With Sickle Cell Disease
Brief Title: Methylphenidate to Address Attention and Executive Deficits Among Children With Sickle Cell Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARS
Record Dates: First submitted 2025-10-22; First posted 2025-11-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease; Executive Dysfunction; Cognitive Impairment; Attention Deficit/Hyperactivity Disorder (ADHD)
Keywords: SCD; ADHD
MeSH Terms: conditions — Anemia, Sickle Cell; Cognitive Dysfunction; Attention Deficit Disorder with Hyperactivity | interventions — 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Intervention Model Description: 30 patients + 42 caregivers (including 12 caregivers who declined participation for interviews)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Methylphenidate Treatment Group (Experimental): All participants in this single-arm pilot study will receive extended-release methylphenidate for 4 weeks. The intervention is designed to evaluate feasibility, acceptability, adherence, and safety of stimulant treatment in children and adolescents with sickle cell disease (SCD) and executive functioning deficits.
  Interventions: Drug: Extended-Release Methylphenidate

INTERVENTIONS:
Drug: Extended-Release Methylphenidate — Participants will receive a weight-based dose of extended-release methylphenidate (0.6 mg/kg/day), rounded to either 10 mg or 20 mg, taken orally once daily for 4 weeks.
  Other Names: MPH

SUMMARY:
The purpose of this study is to determine if patients with sickle cell disease (SCD) can consistently take a drug called Methylphenidate (MPH) daily, once a day for 4 weeks to help with any thinking, attention or schoolwork problems and if they have any side effects.

The study will assess any thinking or attention problems participants may have both before taking this drug and after. Additionally, the study will assess the decision-making process of the caregiver that may influence using this drug or not.

Primary Objective:

• Assess the feasibility, acceptability, and adherence to MPH treatment in children with SCD and EF deficits.

Secondary Objective:

• Evaluate neurobehavioral and safety outcomes following MPH treatment.

Exploratory Objective:

• Evaluate decision-making and determinants influencing methylphenidate utilization among parents.

DETAILED DESCRIPTION:
Children with sickle cell disease (SCD) are at higher risk for executive functioning (EF) deficits, including attention, working memory, and inhibitory control. These deficits are associated with poor academic performance, reduced quality of life, and challenges transitioning to adult healthcare. Despite the effectiveness of stimulant medications like methylphenidate (MPH) in improving EF in the general population and other medical groups, their use in children with SCD is rare.

This is a single-arm, open-label pilot trial conducted at St. Jude Children's Research Hospital. Thirty children with SCD and EF deficits will receive a 4-week course of extended-release MPH (10 mg or 20 mg daily, based on weight). Extended-release methylphenidate will be administered once daily for 4 weeks. The initial dose will be given in clinic, followed by home administration. Adherence will be monitored via weekly video pill counts.

The study will enroll 30 patients aged 8.0 to 17.9 years with SCD and EF impairment, along with 30 caregivers. An additional 12 caregivers who decline participation will be interviewed to assess decision-making and treatment barriers.

Neurobehavioral assessments and side effect evaluations will be conducted at baseline, immediately post-dose, and weekly during the home medication phase. Parents will complete rating scales and interviews to assess treatment acceptability and decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SCD of any genotype
* Enrolled on the institutional protocol: Sickle Cell Clinical Research Intervention Program (SCCRIP)
* Between the ages of 8.0 and 17.9 years

  *Included if performance measure or rating scale criteria met:
* *Score below the 16th percentile on any 2 out of 4 performance measures:

  * NIH Toolbox Flanker
  * NIH Toolbox List Sorting
  * NIH Toolbox Dimensional Change Card Sort Test (DCST)
  * Wechsler Intelligence Scale for Children (WISC) -5/ Wechsler Adult Intelligence Scale (WAIS)-4 Digit Span Forward (DSF)
* *Score above the 84th percentile on any 1 out of 2 parent rating scales:

  * BRIEF-2 Global Executive
  * BASC-3 Attention
* English as the primary language
* Research participant and one parent willing to participate and provide consent/assent according to institutional guidelines
* Negative pregnancy test

Exclusion Criteria:

* Primary language other than English
* Score below the 2nd percentile on the Wechsler Abbreviated Scale of Intelligence (WASI)-2 intelligence quotient (IQ) test
* Uncontrolled seizures (seizure within the past 6 months)
* Cardiomyopathy or known congenital structural cardiac defects
* Stenotic valvular disease, left coronary artery stenosis, or history of myocarditis or pericarditis
* History of heart arrhythmia including ventricular tachycardia, ventricular fibrillation, supraventricular tachycardia, QT prolongation or concomitant use of medications associated with QT prolongation
* Two or more prior episodes of priapism
* Uncontrolled or untreated hypertension
* Stimulant medication within the past two weeks
* Severe sensory loss
* Previous adverse reaction to methylphenidate
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Currently prescribed another investigational medication.
* Currently prescribed any of the following:

  * Phenobarbital (anticonvulsant)
  * Phenytoin (anticonvulsant)
  * Primidone (anticonvulsant)
  * Warfarin (anticoagulant)
  * Antipsychotic medications
  * Selective Serotonin Reuptake Inhibitor (SSRI) medications
  * Tricyclic antidepressant (TCA) medications
  * Vasopressor medications

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Assess feasibility of methylphenidate | Feasibility is measured during the initial recruitment process for each participant.
  Feasibility is measured by the participation rate (i.e., ratio of those who agree to participate to those approached).
Assess acceptability of methylphenidate | Acceptability ratings are captured at baseline and after 4 weeks of treatment with methylphenidate.
  Acceptability is captured by parent- and self-report ratings on the Acceptability of Intervention Measure (AIM).
Assess adherence to methylphenidate | Adherence is measured on a weekly basis through 4 weeks of treatment
  Adherence is measured through weekly pill counts. The primary adherence outcome is the ratio of the number of pills taken to those dispersed.

SECONDARY OUTCOMES:
Behavior Assessment System for Children, 3rd Edition (BASC-3), Parent Report | Baseline and 4-6 weeks after treatment
  Attention, Hyperactivity, and Depression scales are calculated. The investigators will determine the amount and pattern of missing data. The relative change (defined as (post - pre)/pre)) will be calculated for each outcome and rank these changes to determine sensitivity of the measures. The goal of measuring neurobehavioral outcomes in this pilot trial is to determine how feasible the measures are for the target population and their relative sensitivity to the effects of methylphenidate treatment.
Behavior Rating Inventory of Executive Function, 2nd Edition (BRIEF-2), Parent Report | Baseline and 4-6 weeks after treatment
  Global Executive Composite Scale is calculated. The investigator will determine the amount and pattern of missing data for neurobehavioral outcomes. The relative change (defined as (post - pre)/pre)) will be calculated for each outcome and rank these changes to determine sensitivity of the measures. The goal of measuring neurobehavioral outcomes in this pilot trial is to determine how feasible the measures are for the target population and their relative sensitivity to the effects of methylphenidate treatment.
Pediatric Quality of Life Inventory (PedsQL) Sickle Cell Disease modules, Parent Report | Baseline and 4-6 weeks after treatment
  The investigator will determine the amount and pattern of missing data for neurobehavioral outcomes. The relative change (defined as (post - pre)/pre)) will be calculated for each outcome and rank these changes to determine sensitivity of the measures. The goal of measuring neurobehavioral outcomes in this pilot trial is to determine how feasible the measures are for the target population and their relative sensitivity to the effects of methylphenidate treatment.
Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue modules, Parent Report | Baseline and 4-6 weeks after treatment
  The investigator will determine the amount and pattern of missing data for neurobehavioral outcomes. The relative change (defined as (post - pre)/pre)) will be calculated for each outcome and rank these changes to determine sensitivity of the measures. The goal of measuring neurobehavioral outcomes in this pilot trial is to determine how feasible the measures are for the target population and their relative sensitivity to the effects of methylphenidate treatment.
Conners 4th Edition Short Form, Self Report | Baseline and 4-6 weeks after treatment
  The investigator will determine the amount and pattern of missing data for neurobehavioral outcomes. The relative change (defined as (post - pre)/pre)) will be calculated for each outcome and rank these changes to determine sensitivity of the measures. The goal of measuring neurobehavioral outcomes in this pilot trial is to determine how feasible the measures are for the target population and their relative sensitivity to the effects of methylphenidate treatment.
NIH Toolbox Cognition | Baseline and ~90 minutes after first dose administered
  Dimensional Change Card Cort, Flanker, Pattern Comparison, Picture Sequence Memory Test, Picture Vocabulary subtests are completed. The investigator will determine the amount and pattern of missing data for neurobehavioral outcomes. The relative change (defined as (post - pre)/pre)) will be calculated for each outcome and rank these changes to determine sensitivity of the measures. The goal of measuring neurobehavioral outcomes in this pilot trial is to determine how feasible the measures are for the target population and their relative sensitivity to the effects of methylphenidate treatment.
Woodcock Johnson Tests of Academic Achievement, 4th Edition (WJ-IV) | Baseline and ~90 minutes after first dose administered
  Math Fluency subtest is completed. The investigator will determine the amount and pattern of missing data for neurobehavioral outcomes. The relative change (defined as (post - pre)/pre)) will be calculated for each outcome and rank these changes to determine sensitivity of the measures. The goal of measuring neurobehavioral outcomes in this pilot trial is to determine how feasible the measures are for the target population and their relative sensitivity to the effects of methylphenidate treatment.
Measure key safety outcomes using the Side Effects Rating Scale (SERS) | Baseline in-clinic assessments followed by remote weekly assessments for 4 weeks
  The investigator will record all adverse effects reported by participants and categorize adverse effects by type and severity based on the Side Effects Rating Scale. The investigator will present summary statistics, including the number of participants experiencing each type of adverse effect, the severity and the overall percentage of participants affected.
Measure key safety outcomes using the Systematic Assessment for Treatment Emergent Effects | Baseline in-clinic assessments followed by remote weekly assessments for 4 weeks
  The investigator will record all adverse effects reported by participants and categorize adverse effects by type and severity based on the Systematic Assessment for Treatment Emergent Effects. The investigator will present summary statistics, including the number of participants experiencing each type of adverse effect, the severity, and the overall percentage of participants affected

OTHER OUTCOMES:
Evaluate decision-making and determinants influencing methylphenidate utilization among parents | Baseline and 4-6 weeks after treatment
  Semi-structured interviews will be conducted. The interviews will be transcribed and qualitatively coded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Heitzer, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols